CLINICAL TRIAL: NCT06535646
Title: MITO-VATION - Feasibility of a Technology-supported Structured Home Exercise Program in Mitochondrial Disease?
Brief Title: Digital Health Technology for People With Mitochondrial Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Neuroscience Research Australia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2024_ETH00250
Record Dates: First submitted 2024-07-11; First posted 2024-08-02 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Mitochondrial Diseases
MeSH Terms: conditions — Mitochondrial Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Home exercise program (Experimental): All participants will be remotely monitored for 8-weeks, provided with a customised, structured home exercise program and activity monitor smart watch. Training volume will increase gradually. Participants will receive weekly, individualised emails supporting their exercise program, weekly telehealth coaching sessions and pre-programmed smart watch movement reminders.
  Interventions: Other: Home exercise program using Physitrack exercise program and a smart watch

INTERVENTIONS:
Other: Home exercise program using Physitrack exercise program and a smart watch — Participants wear a smart watch to monitor activity levels while using a web based exercise program to follow along for 8 weeks.

SUMMARY:
Abstract: A lack of exercise combined with low levels of activity is prominent in people with Mitochondrial Disease (MD). Unfortunately, access to health professionals such as physiotherapists with experience in MD is difficult, especially in remote areas. The use of digital health technology (DHT) may be a feasible and acceptable way to remove access barriers while increasing participant compliance and self-efficacy with exercise. Given that the implementation of DHT to improve exercise compliance is scalable and inexpensive, it's important to test this intervention clinically. Objective: To determine the feasibility and acceptability of a structured home exercise program, supported by DHT, in people with MD. Methodology: Ten to 15 participants from the MD clinic at Neuroscience Research Australia will be recruited for this study. All participants will be remotely monitored for 8-weeks, provided with a customised, structured home exercise program and activity monitor smart watch. Training volume will increase gradually. Participants will receive weekly, individualised emails supporting their exercise program, weekly telehealth coaching sessions and pre-programmed smart watch movement reminders. Physical performance measures will be taken at week 0, pre-intervention and week 9, post-intervention. Questionnaires on fatigue, quality of life and acceptability of the program will also be administered. Results: Feasibility will be determined from the percentage of participants who enrol in the study from the eligible pool, percentage of dropouts over the study duration, and the percentage who adhere to the exercise program (defined as completing ≥75% of the regimen). Acceptability outcomes will be extracted from post-program questionnaires. Descriptive statistics of outcome measures (means and standard deviations) and any changes from pre to post will also be calculated. Conclusion: If shown to be feasible and acceptable, this intervention has the potential to deliver a significant impact on the lives of individuals with MD and the wider MD community.

DETAILED DESCRIPTION:
Feasibility study

Baseline measurements taken at: week 0 = pre-intervention, Outcome measurements taken at: week 9 = post-intervention assessment

Feasibility outcomes:

1. the percentage of participants who enrol in the study from the eligible pool
2. percentage of dropouts over the study duration
3. Compliance to the exercise program and use of DHT:

   * daily step count goal met from Garmin smart watch data over 56 days expressed as a percentage.
   * weekly intensity minute's goal met from Garmin smart watch over 8 weeks expressed as a percentage.
   * Strength training adherence (from exercise diary) expressed as a percentage of the prescription (3 sessions per week over 8 weeks or 24 planned sessions).
   * Participation in telehealth sessions, expressed as a percentage of the overall prescription (8 telehealth sessions over the 8-week intervention).
   * Wearing of the smart watch (Garmin) for 8 consecutive weeks (56 days), expressed as a percentage of total wear time (24 hours a day, 7 days a week (excluding showering and recharging of device).

Compliance is defined as having met 75% or greater of prescribed activity. Acceptability outcomes will be extracted from post-program questionnaires.

Secondary outcomes:

* 10 Meter Walking Speed - assesses walking speed in meters per second over a short duration.
* 6-Minute Walk Test - walking endurance, distance walked in meters over 6 minutes.
* 5 Time Sit to Stand - lower limb strength, time in seconds taken to perform 5 sit to stands from a standard height chair (43 to 45cm).
* Grip Strength - hand isometric grip strength contraction held for 3-5 seconds, measuring grip strength in kilograms.
* Berg Balance Test - 14-item scale designed to measure balance, scored out of 56.
* Fatigue Impact Scale - self-reported questionnaire evaluating the effect of fatigue on three domains of daily life: cognitive functioning, physical functioning, and psychosocial functioning, 40 items, each scored 0 (no problem) to 4 (extreme problem), providing a continuous scale of 0-160.
* Newcastle Mitochondrial Disease Adult Scale - rating scale to monitor the progression of a PMD. Sections 1 & 2 are self-rated while section 3 is rated by a neurologist.

Home Exercise Program All participants will be provided with a structured home exercise program which is customised according to the participant's baseline activity measures obtained from smart watch data over 1 week pre-intervention (week 0). This home exercise program is undertaken using the supplied smart watch (Garmin), Physitrack app and elastic bands. An education session on how to use the training equipment will be conducted week 1- start of intervention appointment at Neuroscience Research Australia (NeuRA). A narrated video of the exercise program will also be sent to participants via email through the Physitrack app. A hard copy version of the exercise program will be supplied to participants along with an exercise diary at the week 1 start of intervention appointment.

The home exercise intervention will last 8 weeks and consist of:

1. A daily step target goal.
2. A weekly intensity minutes target goal.
3. Major muscle group strengthening using the supplied equipment.

Daily step target:

Participants will attempt to increase their daily step count by 10% each week from baseline, until an increase of 50% is achieved at week 5. This volume will be then maintained or increased as tolerated for the remaining 3 weeks until the intervention ends. The means by which daily step count is achieved is up to the participant (i.e. planned walk or increased habitual walking activity). Participants will be able to view live on their smart watch or via Garmin Connect app, how many steps they have taken at any time to help them meet their daily step target.

Intensity minutes target goal:

Intensity minutes are earned based on a participant's current heart rate when compared to their average resting heart rate. Intensity minutes are earned once increased activity is detected by the smart watch. Participant's age, weight, height, and resting heart rate calculated by the Garmin device also factor into intensity minutes. Participants will attempt to increase their weekly intensity minutes score by 10% each week from baseline, until an increase of 50% is achieved at week 5. This volume will be then maintained or increased as tolerated for the remaining 3 weeks until the intervention ends.

Strength training:

Each home strength training session (3 per week) will start with a short warm up, i.e. 5-min walk to be followed by 6 stretching exercises targeting the lower limb, upper limb and spine.

Once warmed up, participants will perform a circuit of 8 exercises with the help of the Physitrack app or hard-copy exercise program. It will involve large muscle groups in the following order (i.e. alternating arm and leg exercises to minimise muscle soreness and fatigue):

1. Lunges
2. Row
3. Sit to stand
4. Chest press
5. Hip abduction
6. Trunk rotation
7. Hip extension
8. Heel raise

Sets and repetitions for each participant, along with training intensity (i.e., elastic band resistance) will be determined using pre-intervention assessment baseline data during the face-to-face meeting at the beginning of week 1. The modified Borg rating of perceived exertion scale (1 to 10) will be used where a score of 6 (i.e. able to speak 3 to 5 words comfortably) being the starting level. Once a score of 5 (i.e. able to speak more than 5 words comfortably) or less is perceived, the band resistance will be raised to the next level. The circuit of 8 exercises will consist of 1 to 3 rounds of single sets (10 to 20 repetitions) to allow full muscle group recovery in between. The speed of repetitions will focus on having a controlled concentric/eccentric portion of the movement. The training volume (sets x reps x band resistance) will be increased by 10% per week for 5 weeks and then maintained or increased as tolerated for a further 3 weeks. The volume targets will be emailed to participants weekly through the Physitrack app. Targets will also be discussed at the weekly telehealth session.

Participants will complete a supplied daily exercise diary for monitoring of adherence to the prescribed exercise program.

Telehealth coaching sessions

Eight, weekly telehealth meetings will take place at a time that is suitable for the study participant, starting week 1 and continue through to week 8 of the study. Each session will last 10 to 20 minutes via phone using the Physi app or through an email link to a home computer. The aim of each meeting will be to monitor participant progress and troubleshoot any barriers or unforeseen difficulties that may arise across the week to maintain motivation for exercise. Health coaching strategies will be used such as:

* use of a health coaching log form
* setting clear goals
* establishing a trusting relationship
* using active listening and questioning techniques
* providing constructive feedback
* support to encourage independence in exercising
* adaptability and flexibility to tailor the session to meet the needs and preferences of each individual participant In instances where technical difficulties prevent a participant from being able to log in to a telehealth session it may still be conducted over the phone.

Physitrack health coaching email messages Physitrack is an exercise prescription app which allows remote contact between therapist's and their patients. Participants will need to download the Physitrack app onto their phones to be able to receive weekly emails and participate in weekly telehealth meetings. Personalised emails will be sent from Physitrack to participants at the beginning of each week and consist of encouraging messages and reminders of the benefits of exercise. They will also include fully narrated exercise videos so participants will have a clear understanding of their exercise program and goals each week. They will be scheduled to be sent to the participant's email each Monday morning between weeks 2 and 8 of the study. In the case of week 1, the email will be sent after the activity data has been downloaded and reviewed by the investigator at the week 1 start of intervention meeting that will occur in-person.

Activity monitoring

All participants will have their activity monitored 24 hours a day, 7 days a week (excluding showering and device recharging) for 8 weeks using a smart watch (Garmin). The smart watch will record activity during and outside of the personalised home exercise program. Participants will be provided with the smart watch at the conclusion of the pre-intervention meeting (week 0), to wear for one week to determine baseline activity levels. This data will be downloaded at the study visits at the beginning of week 1 (start of intervention meeting) and post-intervention assessment at the beginning of week 9. Participants will download the Garmin Connect app onto their smartphone and transfer data daily to avoid any potential loss of information. The metrics downloaded will include:

* Steps taken per day
* Average heart rate
* Intensity minutes
* Hours of sleep per day

A brief (5 minute) training session will be held at the end of the pre-intervention visit to teach the participants how to wear, charge, and operate the smart watch. A more detailed training session will be held at the week 1 start-intervention visit to NeuRA. Participants will be taught how to use the smart watch and Garmin Connect app to self-monitor their daily activity levels and work toward meeting their daily and weekly activity goals.

STUDY GROUPS

Single group pre-post feasibility study. Participants will be those with a primary diagnosis of PMD who attend the PMD clinic at Neuroscience Research Australia (NeuRA). Participants will attend 3 study appointments at the following time points:

* Pre-intervention - week 0, for initial assessment of baseline objective and subjective measures, provision of a smart watch (Garmin), education on its use and downloading of the Garmin Connect app onto participants phones. The watch is worn continuously for 1 week before returning for the next face to face meeting where baseline activity data will be downloaded for review.
* Start-intervention - beginning of week 1, for downloading of 1 week of pre-intervention activity data to set exercise targets. Education on performing the prescribed home exercise program including use of supplied equipment (smart watch, elastic bands & exercise diary). The home exercise program will be provided both electronically using the Physitrack app downloaded onto participants phones and in hard copy via an exercise diary for participants to fill in as required.
* Post-intervention - beginning of week 9, for reassessment of measures conducted at the pre-intervention assessment week 0. Downloading of 8 weeks of participant activity data from their Garmin Connect app. Gain feedback on program acceptability from participants via questionnaires which will contain questions regarding the home exercise experience, smart watch, telehealth and Physitrack use.

NUMBER OF PARTICIPANTS This study will recruit 10 participants with a PMD over a 5-month period.

NUMBER OF CENTRES

* This study will be conducted at a single site, NeuRA, Randwick, NSW.
* This study will be completed over a 1-year period: 5-months recruitment, a 5-month trial period and 2-months to analyse and report the results. The expected start date is July 2024.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Have a confirmed diagnosis of a PMD
* Be able to walk a minimum of 6 minutes with or without rest
* Provide written informed consent and
* Willingness and ability to comply with the study procedures
* Own a smart phone and be willing to download 2 apps
* internet access/telehealth app

Exclusion Criteria:

* Have atrial fibrillation or untreated symptomatic cardiac arrhythmia
* Non-English speaking
* Are pregnant
* Are wheelchair bound
* Have visual acuity less than 6/60 (Snellen Test)
* Other co-morbidities such as severe osteoarthritis, balance impairment, chronic obstructive pulmonary disease, cognitive impairment, depression and anything else that would impact on participant adherence, participant safety or interpretation of results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-09-09 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Feasibility - recruitment rate | 8 weeks
  A recruitment rate of at least 50% of the people screened will be deemed feasible.
Feasibility - retention rate | 8 weeks
  A retention rate of 80% of participants will be deemed feasible.
Feasibility - adherence to the exercise intervention | 8 weeks
  An adherence to the exercise intervention is set at 75% to be deemed feasible.
Acceptability of platforms used | 8 weeks
  Acceptability subjective questionnaires will explore the intervention in terms of instructions given, useability and desirability of platforms used.

SECONDARY OUTCOMES:
Physical performance test 1 | 8 weeks
  10 Meter Walking Speed - meters per second.
Physical performance test 2 | 8 weeks
  6-Minute Walk Test - distance walked in 6 minutes measured in meters over a 20 meter course.
Physical performance test 3 | 8 weeks
  5 Time Sit to Stand - time in seconds taken to perform 5 sit to stands from a standard height chair.
Physical performance test 4 | 8 weeks
  Grip Strength - isometric grip strength of both hands measured in kilograms.
Physical performance test 5 | 8 weeks
  Berg Balance Test - 14-item scale measuring balance. Scored on a 5-point ordinal scale ranging from 0 to 4, with 0 indicating an inability to complete the task entirely and 4 indicating an ability to complete the task criterion. A high score correlates to better balance.
Subjective measure 1 | 8 weeks
  Fatigue Impact Scale - self-reported questionnaire on fatigue, 40 items, each scored 0 (no problem) to 4 (extreme problem), providing a continuous scale of 0-160. A high score equates to greater fatigue.
Subjective measure 2 | 8 weeks
  Newcastle Mitochondrial Disease Adult Scale - monitors disease progression Section 1 - rates current function according to the patient, 10 questions rated 0 to 5 with 0 being normal and 5 unable to do.
  Section 2 - this 9 item section rates system specific involvement from 0 (no past history) to 5 (significant history) according to the patient interview, clinician's knowledge of the patient and the clinical notes.
  Section 3 - rates the patient's current status according to the examination performed by the rater. Scores are assigned according to the clinician's judgement. This 10 question section is rated 0 to 5 with 0 being none and 5 being severe.
  A final total score is calculated by simply summing the scores obtained for each section. The higher the score the more severe the disease. Total scores can range from 0 to 145.

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn M Sue, MBBS, PhD, FRACP, Principal Investigator — Professor and Director, Kinghorn Chair, Neurodegeneration at NeuRA and Director of Neurosciences at POWH
Locations (1):
- Neuroscience Research Australia, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No